CLINICAL TRIAL: NCT02749149
Title: Assessment of the Frailty Score in Cardiac Surgery and Its Correlation to Cardiac Postoperative Morbidity and Disability - a Prospective Observational Study
Brief Title: Does Frailty Help Predict Postoperative Outcomes in Cardiac Surgery?
Acronym: FOCuS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH16-012
Record Dates: First submitted 2016-04-08; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Heart Disease; Heart Valve Diseases
Keywords: Cardiac; Surgery; Frailty; Frail; Patients; Recovery; Morbidity; Outcomes; Mortality; Heart; Perioperative; Disability; WHODAS
MeSH Terms: conditions — Coronary Disease; Heart Valve Diseases; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac Surgery: Patients undergoing cardiac surgery: coronary artery bypass graft (CABG); valve replacement/repair; or transcatheter aortic valve implantation (TAVI) surgery

SUMMARY:
This study will assess the benefit in using a frailty score to quantify accurate risk pre-operatively in patients undergoing major cardiac surgery in order to predict morbidity and disability-free survival post-operatively.

DETAILED DESCRIPTION:
Increasingly, the group of patients undergoing cardiac surgery are older. Patients that are more elderly and frail are known to have an increase risk of injury to major organs following surgery including the heart, kidneys, and brain, all of which are associated with worse survival or diminished quality of life. It is becoming more important to be able to predict how well patients will fair in cardiac surgery, including predicting risk of complications (such as stroke or heart attacks) as well as long-term survival and quality of life. Currently, scores such as EUROscore can be used with good effect in predicting survival and major complications in cardiac surgery patients. However, frailty - the severity of a patient's weakness or fragility - has emerged as a potential candidate in predicting risk. Recent research has shown frailty score to predict risk of survival and complications following cardiac surgery and suggested to be possibly superior to pre-existing scores. The investigators wish to investigate the possible link between frailty and outcomes following cardiac surgery, in addition to current risk scores. The investigators also wish to determine whether frailty can effectively predict longer-term outcomes such as 'disability-free survival' - a patient-centred score that measures the ability of a patient to lead normal life activities. Patients undergoing major cardiac surgery at King's College Hospital will be recruited, following consent. The study will mainly involve questionnaires at various stages, starting at a pre-operative clinic. After surgery, follow up of patient's progress will be carried out at 3 days in hospital; and at 1 month, 3 months, and 6 months and 1 year via telephone. The investigators expect the results of this observational study to influence further research into the use of frailty risk scoring prior to clinical decisions, and add to the evidence in assessing risk-related outcomes in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Due to undergo elective cardiac surgery: coronary artery bypass graft (CABG); valve replacement/repair; or transcatheter aortic valve implantation (TAVI) surgery
* Able to give informed consent
* Fluency in English

Exclusion Criteria:

* Emergency cardiac surgery and non-cardiac surgery
* Inadequate knowledge of English that will prevent patients from completing the consent or undertaking study assessments
* Severe visual, auditory, or motor handicap
* Concurrent diseases of the central nervous system,
* Patients at the extremes of frailty, in whom it would be unethical to perform a full assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators are planning to recruit 120 adult patients undergoing elective coronary artery bypass graft (CABG); valve replacement/repair; or transcatheter aortic valve implantation (TAVI) surgery at King's College Hospital, Denmark Hill, London
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Disability-free survival | 1 year
  Defined as percentage of participants alive and with a disability score (using World Health Organisation Disability Assessment Schedule 2.0, WHODAS) of less than 25%.

SECONDARY OUTCOMES:
Mortality | 1 month postoperative
Delirium | 3 days postoperative
  Using Confusion Assessment Method (CAM).
In hospital complications | 1 month
  Incidence of major adverse cardiac or cerebrovascular events, and/or acute renal injury.
Return to theatre | 1 month
Length of hospital stay | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lucas de Carvalho, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: No
Contact research lead.